CLINICAL TRIAL: NCT06703203
Title: A Single-center, Randomized, Double-blind, Active-controlled Phase I/II Clinical Trial to Evaluate the Safety and Immunogenicity of 26-valent Pneumococcal Conjugate Vaccine in People Aged 2 Months and Older
Brief Title: Phase I/II Clinical Trial of 26-valent Pneumococcal Conjugate Vaccine
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beijing Zhifei Lvzhu Biopharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 202417AB
Record Dates: First submitted 2024-11-21; First posted 2024-11-25 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Pneumococcal Vaccines
Keywords: 26 valent pneumococcal conjugate vaccine
MeSH Terms: interventions — 23-valent pneumococcal capsular polysaccharide vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- ≥60 years old age group (for phase Ⅰ) (Other): There are 30 subjects in ≥60 years old age group, randomly assigned to the experimental group and the control group in a 2:1 ratio.
  Interventions: Biological: 26-Valent pneumococcal conjugate vaccine; Biological: 23-Valent pneumococcal polysaccharide vaccine
- 18-59 years old age group (for phase Ⅰ) (Other): There are total 40 subjects in 18-59 age group. Among them, 30 subjects were randomly assigned to the experimental group and the control group in a 2:1 ratio. In addition, other 10 subjects aged 18-55 to receive the experimental vaccine as the serum calibration test population.
  Interventions: Biological: 26-Valent pneumococcal conjugate vaccine; Biological: 23-Valent pneumococcal polysaccharide vaccine
- 6-17 years old age group (for phase Ⅰ) (Other): There are 30 subjects in 6-17 years old age group, randomly assigned to the experimental group and the control group in a 2:1 ratio.
  Interventions: Biological: 26-Valent pneumococcal conjugate vaccine; Biological: 23-Valent pneumococcal polysaccharide vaccine
- 2-5 years old age group (for phase Ⅰ/Ⅱ) (Other): There are total 230 people in 2-5 years old age group. Among them, there were 30 subjects included in the phase Ⅰ clinical trial and were randomly assigned to the experimental group and the control group in a 2:1 ratio. And the other 200 people were included for phase Ⅱ and were randomly assigned to the experimental group and the control group in a 1:1 ratio.
  Interventions: Biological: 26-Valent pneumococcal conjugate vaccine; Biological: 13-Valent pneumococcal conjugate vaccine
- 13-23 months old age group (for phase Ⅰ) (Other): There are 30 subjects in 13-23 months old age group, randomly assigned to the experimental group and the control group in a 2:1 ratio.
  Interventions: Biological: 26-Valent pneumococcal conjugate vaccine; Biological: 13-Valent pneumococcal conjugate vaccine
- 7-11 months old age group (for phase Ⅰ) (Other): There are 30 subjects in 7-11 months old age group, randomly assigned to the experimental group and the control group in a 2:1 ratio.
  Interventions: Biological: 26-Valent pneumococcal conjugate vaccine; Biological: 13-Valent pneumococcal conjugate vaccine
- 3 months old age group (for phase Ⅰ) (Other): There are 30 subjects in 3 months old age group, randomly assigned to the experimental group and the control group in a 2:1 ratio.
  Interventions: Biological: 26-Valent pneumococcal conjugate vaccine; Biological: 13-Valent pneumococcal conjugate vaccine
- 2 months old age group （for phase Ⅰ） (Other): There are 30 subjects in 2 months old age group, randomly assigned to the experimental group and the control group in a 2:1 ratio.
  Interventions: Biological: 26-Valent pneumococcal conjugate vaccine; Biological: 13-Valent pneumococcal conjugate vaccine

INTERVENTIONS:
Biological: 26-Valent pneumococcal conjugate vaccine — As an experimental group. The active ingredient of 26-valent pneumococcal conjugate vaccine is the capsular polysaccharide of 26 pneumococcal serotypes conjugated to the tetanus toxoid carrier protein. Administer one dose of 0.5mL each time.
Biological: 23-Valent pneumococcal polysaccharide vaccine — As a control group. The effective ingredients of 23-valent pneumococcal polysaccharide vaccine are 23 serotypes of pneumococcal capsular polysaccharides. Administer one dose of 0.5mL each time.
  Arms: 18-59 years old age group (for phase Ⅰ); 6-17 years old age group (for phase Ⅰ); ≥60 years old age group (for phase Ⅰ)
Biological: 13-Valent pneumococcal conjugate vaccine — As a control group. The active ingredient of 13-valent pneumococcal conjugate vaccine is the capsular polysaccharide of 13 pneumococcal serotypes conjugated to the tetanus toxoid carrier protein. Administer one dose of 0.5mL each time.
  Arms: 13-23 months old age group (for phase Ⅰ); 2 months old age group （for phase Ⅰ）; 2-5 years old age group (for phase Ⅰ/Ⅱ); 3 months old age group (for phase Ⅰ); 7-11 months old age group (for phase Ⅰ)

SUMMARY:
The purpose of this experiment is to evaluate the safety and immunogenicity of the 26 valent pneumococcal conjugate vaccine in the population aged 2 months and above.

DETAILED DESCRIPTION:
A single-center, randomized, double-blind, active-controlled trial design (Phase I/II) was used. In addition, according to the requirements in the approval letter of this product (2024LP01053), serum standards need to be established for the newly added types (24F, 35B). Therefore, a calibration group is set and an open study design is adopted.

ELIGIBILITY:
Inclusion Criteria:

* The subject is 2-3 months old (minimum 6 weeks old), 7 months old and above at the time of enrollment, and the legal guardian and/or the subject can provide legal identification certificate;
* The subjects themselves and/or their legal guardians understand the vaccination and trial procedures, voluntarily participate in the trial and sign the informed consent form;
* The subject and/or legal guardian can comply with the clinical trial protocol, have the ability to use thermometer, scale and fill in diary card and contact card as required;
* Female subjects of childbearing potential agree to take effective contraceptive measures from enrollment to 6 months after vaccination.
* For calibration group subjects: 18 to 55 years of age, ≥ 50 kg for males or ≥ 45 kg for females.

Exclusion Criteria:

* Axillary body temperature ≥ 37.3 ℃ on the day of enrollment;
* History of infectious diseases caused by Streptococcus pneumoniae confirmed by bacterial culture within 3 years;
* Have received or plan to receive a Streptococcus pneumoniae vaccine outside the trial protocol, including marketed or other investigational Streptococcus pneumoniae vaccines;
* Pregnant or lactating women; Previous history of severe allergy to any vaccine or drug, such as urticaria, dyspnea, angioneurotic edema, anaphylactic shock, Henoch-Schonlein purpura, thrombocytopenic purpura;
* Allergic to any component of the investigational vaccine;
* Suffering from severe respiratory diseases (such as severe asthma), heart diseases, liver diseases, kidney diseases, congenital malformations, developmental disorders and genetic defects (including but not limited to: down syndrome, thalassemia major, etc.) that may interfere with the conduct or completion of the trial;
* Diagnosed with congenital or acquired immunodeficiency, or suspected to have serious chronic disease or systemic disease that may interfere with the conduct or completion of the trial, such as: active tuberculosis, human immunodeficiency virus (HIV) infection, etc.;
* Encephalopathy, uncontrolled epilepsy, convulsion and other progressive neurological diseases, or a history or family history of mental illness;
* Contraindications for intramuscular injection such as thrombocytopenia, any coagulation disorder or receiving anticoagulant therapy;
* Asplenia or splenectomy, functional asplenia due to any condition;
* Immunosuppressant therapy, cytotoxic therapy or corticosteroid therapy within 3 months prior to vaccination, such as systemic glucocorticoid therapy for more than 2 consecutive weeks, such as prednisone or similar drugs > 5 mg/day (excluding corticosteroid spray therapy for allergic rhinitis, surface corticosteroid therapy for acute non-complicated dermatitis);
* Received blood products or immunoglobulins within 3 months prior to enrollment (hepatitis B immunoglobulin is acceptable), or planned to be used during the trial (before the last immunogenicity blood sample collection);
* Within 3 days before the first dose of vaccine, the patient has acute illness or is in acute attack of chronic disease, or has used antipyretic, analgesic or anti-allergic drugs (such as: acetaminophen, ibuprofen, aspirin, etc.);
* Received non-live vaccine within 7 days (≤ 7 days) or live attenuated vaccine within 14 days (≤ 14 days) prior to enrollment;
* Hypertension (systolic blood pressure ≥ 140 mmHg and/or diastolic blood pressure ≥ 90 mmHg, applicable to adults);
* Abnormal and clinically significant laboratory test results, which are not suitable for enrollment as determined by the investigator (applicable to subjects aged 2 years and older in Phase I);
* Birth weight < 2.5 kg, premature delivery (gestational age < 37 weeks), history of abnormal labor process, history of asphyxia rescue, history of nerve organ damage, history of pathological jaundice confirmed by diagnosis;
* For Standardised Subjects:

  ① Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 50 U/L; Or hemoglobin ≤ 115 g/L (female)/120g/L (male); Any positive serology for hepatitis B, hepatitis C, HIV, or syphilis.
* Plans to move before the end of the trial or leave the area for an extended period of time during scheduled trial visits;
* Ongoing participation or planning to participate in other clinical trials (vaccines, drugs, medical devices, etc.) in the near future;
* Subject has any condition that, in the opinion of the investigator, may interfere with the evaluation of the objectives of the trial.

Min Age: 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2024-08-27 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
AE occurrences within 0-30 days after each dose of vaccination (for phase Ⅰ/Ⅱ） | 30 day after each vaccination
  All AE occurrences within 0-30 days after each dose of vaccination (number of cases, incidence rate, and relationship with vaccination)
Solicited AE occurrences within 0-30 minutes after each dose of vaccination (for phase Ⅰ/Ⅱ） | 30 minutes after each vaccination
  The occurrence of Solicited adverse events (AE) within 0-30 minutes after each dose of vaccination (number of cases, incidence rate, and relationship with vaccination)
Solicited AE occurrences within 0-7 days after each dose of vaccination (for phase Ⅰ/Ⅱ） | 0-7 days after each vaccination
  The occurrence of solicited adverse events (AE) within 0-7 days after each dose of vaccination (number of cases, incidence rate, and relationship with vaccination);
Unsolicited AE occurrences within 0-30 days after each dose of vaccination (for phase Ⅰ/Ⅱ） | 0-30 days after each vaccination
  The occurrence of unsolicited adverse events (AE) within 0-30 days after each dose of vaccination (number of cases, incidence rate, and relationship with vaccination);
Grade 3 and above AE occurrences within 0-30 days after each dose of vaccination (for phase Ⅰ/Ⅱ） | 0-30 days after each vaccination
  The occurrence of grade 3 and above adverse events within 0-30 days after each dose of vaccination (number of cases, incidence rate, and relationship with vaccination).
All SAE occurrences within 0-6 months after vaccination (for Phase Ⅱ) | 0-6 months after each vaccination
  The occurrence of all serious adverse reactions within 6 months after vaccination (number of cases, incidence rate, and relationship with vaccination)
Positive rate of serotype-specific pneumococcal IgG antibody on the 30th day after immunization in subjects aged 2-5 years （for phase Ⅱ） | 30 day after vaccination
  Proportion of subjects with serotype-specific pneumococcal IgG antibody concentration ≥ 0.35 μg/ml on Day 30 after vaccination in subjects aged 2-5 years

SECONDARY OUTCOMES:
All SAE in the population aged ≥12 months during 0-6 months after vaccination （for phase Ⅰ） | 0-6 months after vaccination
  All SAE in the population aged 12 months and older from the first dose to 6 months after the full course of vaccination
All SAE in the population aged <12 months from the first dose to 6 months after the primary immunization and from the booster to 6 months after the booster（for phase Ⅰ） | From the first dose to 6 months after the primary immunization and from the booster to 6 months after the booster
  All SAE from the first dose to 6 months after the primary immunization and from the booster to 6 months after the booster in the population less than 12 months of age.
Proportion of IgG antibodies ≥ 1.0 µg/mL and GMC results on Day 30 post-immunization（for phase Ⅱ） | 30 day after vaccination
  Proportion of subjects with serotype-specific pneumococcal IgG antibodies ≥ 1.0 µg/mL and GMC results on Day 30 post-immunization in subjects 2 to 5 years of age.

CONTACTS AND LOCATIONS:
Locations (1):
- Henan Provincial Center for Disease Control and Prevention, Shangqiu, Henan, China

IPD SHARING:
Plan to Share IPD: Undecided